CLINICAL TRIAL: NCT05932147
Title: Pilates Exercise Versus Manual Lymphatic Drainage On Axillary Web Syndrome Post Mastectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, ORCHID SABER, Physiotherapist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/003745
Record Dates: First submitted 2023-06-03; First posted 2023-07-06 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-06

CONDITIONS: Mastectomy; Lymphedema
MeSH Terms: conditions — Lymphedema | interventions — Exercise Movement Techniques; Manual Lymphatic Drainage

STUDY DESIGN:
Intervention Model Description: Group A:( Pilates exercise) This group includes 34 patients who have axillary web syndrome received Pilates exercise with traditional physical therapy exercise program (strength, core stability, flexibility, muscle control, posture and breathing). Patients received 3 sessions per week for 8 weeks; time of session is 30 minutes.
  ) Group B: (Manual Lymphatic Drainage) This group includes 34 patients who axillary web syndrome received Manual lymphatic drainage massage with traditional physical therapy exercise program (strength, core stability, flexibility, muscle control, posture and breathing). Patients received 3 sessions per week for 8 weeks; time of session is 30 minutes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pilates group (Experimental): This group includes 34 patients who have axillary web syndrome will receive Pilates exercise with traditional physical therapy exercise program (strength, core stability, flexibility, muscle control, posture and breathing). Patients will receive 3 sessions per week for 9 weeks; time of session is 30 minutes.
  Interventions: Other: Pilates exercise
- Manual lymphatic massage group (Experimental): This group includes 34 patients who axillary web syndrome will receive Manual lymphatic drainage massage with traditional physical therapy exercise program (strength, core stability, flexibility, muscle control, posture and breathing). Patients will receive 3 sessions per week for 9 weeks; time of session is 30 minutes.
  Interventions: Other: Manual lymphatic massage

INTERVENTIONS:
Other: Pilates exercise — 1. Shoulder Abduction with External Rotation exercise
  2. Shoulder bridge exercise
  3. Mermaid sitting exercise.
  4. Standing Pilates mermaid exercise with towel
  5. Rocking exercise
  6. Saw Pilates exercise.
  7. Bird-dog Pilates exercise.
  8. Roll up exercise.
  9. Cobra pose exercise.
  10. Child pose exercise.
  Arms: Pilates group
Other: Manual lymphatic massage — procedures of Manual lymphatic drainage program Things to know about MLD Massage
  * Use only gentle pressure, just enough to see your skin move.
  * Massage should not be painful.
  * Do not rub your skin red.
  * Do massage each day.
  * Repeat each step 5 to 10 times.
  * The massage should take about 15 to 30 minutes.
  Arms: Manual lymphatic massage group

SUMMARY:
1-Subjects: Sixty-eight patients sample size according to G power who have Axillary web syndrome post mastectomy participated in this study. Their ages ranged from 35 to 55 years. The participants selected from learning hospitals (Al kasr Al Ayni hospital and National cancer institute) and randomly distributed into 2 equal groups.

1.1 Design of study: In this study the patients randomly assigned into two equal groups (34 patients for each group) 1.1(a) Group A: (Pilates Exercise)

1.1(b) Group B: (Manual Lymphatic Drainage)

2. Equipment's and Tools: Equipment in this study divided into two main categories: measuring and therapeutic equipment.

2.1. Measuring Equipment:

The following tools are used to assess Range of motion and pain for shoulder joint:

2.1 (a) Measuring and assessment of pain by:

* Visual analogue scale 2.2 (b) Measuring range of motion (ROM) by:
* Electronic Goniometer 2.3 (c) Measuring Disability of the arm, shoulder and hand by:
* DASH questionnaire (Disability of the arm, shoulder and hand). 2.2. Therapeutic Equipment: 1. Pilates exercise 2- Manual lymphatic drainage 3. Procedures of the study:

The procedures of this study are classified into the following:

3.1 Measurement Procedures: All measurements have been taken before treatment (pre) after 9 weeks (post 1) after 9 weeks (post 2).

1.1 (a) Assessment of pain of shoulder joint

• Assessment of upper limb pain using visual analogue scale 3.1(b) Assessment of Range of motion of shoulder joint: By Electronic Goniometer. 3.1 (c) Assessment of Disability of the arm, shoulder and hand The disabilities of the arm, shoulder and hand questionnaire (DASH) 1.2 Therapeutic procedures: 3.2(a) procedures of Pilates exercise program:

1. Shoulder Abduction with External Rotation exercise
2. Shoulder bridge exercise
3. Mermaid sitting exercise.
4. Standing Pilates mermaid exercise with towel
5. Rocking exercise
6. Saw Pilates exercise.
7. Bird-dog Pilates exercise.
8. Roll up exercise.
9. Cobra pose exercise.
10. Child pose exercise.

DETAILED DESCRIPTION:
1-Subjects: Sixty-eight patients sample size according to G power who have Axillary web syndrome post mastectomy participated in this study. Their ages ranged from 35 to 55 years. The participants have been selected from learning hospitals (Al kasr Al Ayni hospital and National cancer institute) and randomly distributed into 2 equal groups.

1.1 Design of study: In this study the patients randomly assigned into two equal groups (34 patients for each group) 1.1(a) Group A: (Pilates Exercise) This group includes 34 patients who have axillary web syndrome received Pilates exercise with traditional physical therapy exercise program (strength, core stability, flexibility, muscle control, posture and breathing). Patients will receive 3 sessions per week for 8 weeks; time of session is 30 minutes.

1.1(b) Group B: (Manual Lymphatic Drainage) This group includes 34 patients who axillary web syndrome received Manual lymphatic drainage massage with traditional physical therapy exercise program (strength, core stability, flexibility, muscle control, posture and breathing). Patients received 3 sessions per week for 8 weeks; time of session is 30 minutes.

2. Equipment's and Tools: Equipment in this study divided into two main categories: measuring and therapeutic equipment.

2.1. Measuring Equipment:

The following tools are used to assess Range of motion and pain for shoulder joint:

2.1 (a) Measuring and assessment of pain by:

* Visual analogue scale 2.2 (b) Measuring range of motion (ROM) by:
* Electronic Goniometer 2.3 (c) Measuring Disability of the arm, shoulder and hand by:
* DASH questionnaire (Disability of the arm, shoulder and hand). 2.2. Therapeutic Equipment: 1. Pilates exercise

Parameters:

* Duration 30 minutes.
* Patient own choice with guidance.
* Suitable equipment chosen for specific situation.
* Measurement and follow up
* Three session per week
* For 9 weeks 2- Manual lymphatic drainage

Parameters:

* Duration 30 minutes.
* Patient own choice with guidance.
* Suitable equipment chosen for specific situation.
* Measurement and follow up
* Three session per week
* For 9 weeks 3. Procedures of the study:

The procedures of this study are classified into the following:

3.1 Measurement Procedures: All measurements have been taken before treatment (pre) after 9 weeks (post 1) after 9 weeks (post 2).

1.1 (a) Assessment of pain of shoulder joint

* Assessment of upper limb pain using visual analogue scale
* VAS will be used to assess the degree of pain intensity subjectively by same subject. This scale consists of 10cm line with the words "No Pain" on the right side.

3.1(b) Assessment of Range of motion of shoulder joint: By Electronic Goniometer.

* A standardized means of measuring and recording and a goniometer is aligned over a joint and with a click of a button the ROM measurement is entered automatically into E-LINK computer software, generating progress reports that can be utilized as definitive outcome measures. Goniometer to obtain goniometric measurements for shoulder flexion, abduction and external rotation will be used.

  * Measuring of shoulder flexion range while patient is in supine position
  * Measuring of shoulder abduction range while patient in sitting or supine position.
  * Measuring of shoulder external rotation range while patient in supine position. 3.1 (c) Assessment of Disability of the arm, shoulder and hand The disabilities of the arm, shoulder and hand questionnaire (DASH)
* The disabilities of the arm, shoulder and hand (DASH) questionnaire is a self-administered region-specific outcome instrument developed as a measure of self-rated upper-extremity disability and symptoms.
* The DASH consists mainly of a 30-item disability/symptom scale, scored 0 (no disability) to 100 1.2 Therapeutic procedures: 3.2(a) procedures of Pilates exercise program:

  1. Shoulder Abduction with External Rotation exercise
  2. Shoulder bridge exercise
  3. Mermaid sitting exercise.
  4. Standing Pilates mermaid exercise with towel
  5. Rocking exercise
  6. Saw Pilates exercise.
  7. Bird-dog Pilates exercise.
  8. Roll up exercise.
  9. Cobra pose exercise.
  10. Child pose exercise.

ELIGIBILITY:
Inclusion Criteria:

* • Age range between 35-55 years.

  * Number of dissection of lymph nodes.
  * No change of arm size.
  * Females only will participate in the study.
  * All patients have axillary web syndrome
  * All patients' relatives enrolled to the study will have their informed consent

Exclusion Criteria:

* • Age more than 55 years or less than 35 years.

  * Lymphedema.
  * Chemotherapy and Radiotherapy.
  * Pregnant women.
  * Patients who suffer from mental or psychological problems.
  * Patients who have psoriasis, liver disease, diabetes mellitus, hypertensive patients and cardiac problems
  * Patients have Genetic disease or deformity
  * Who has previous injury or fracture in shoulder joint
  * Rheumatoid arthritis
  * Osteopenia
  * Frozen shoulder

Ages: 35 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Sixty-eight patients sample size according to G power who have Axillary web syndrome post mastectomy participated in this study.
Enrollment: 68 (Actual)
Dates: Start 2022-07-03 (Actual); Primary Completion 2022-09-04 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Electric Goniometer | 9 weeks
  for RANGE OF MOTION MEASURMENT
DASH SCALE (Disability of arm, shoulder and hand) | 9 weeks
  for disability measurement

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. Haidy N Asham, Study Chair — Professor of Physical Therapy for Surgery; Ass. Prof. Dr. Ereny S Wahba Khalil, Study Director — Assistant professor of Physical Therapy for Surgery; Prof. Dr. Mohamed A Hassan Abolkasem, Principal Investigator — Professor of Clinical Oncology
Locations (1):
- Cairo university of physical therapy, Dokki, Egypt